CLINICAL TRIAL: NCT02196402
Title: Narrow Band Imaging in the Prediction of Surveillance Intervals After Polypectomy in Community Practice: Ready for (a European) Prime Time
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, MD, Valduce Hospital
Other Study IDs: 5/2014
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Resect and Discard Strategies for Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study population: Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy for routine indications (screening, symptoms, surveillance).
  Exclusion criteria:
  * patients with CRC history or hereditary polyposis syndromes or hereditary non-polyposis colorectal cancer
  * patients with inadequate bowel preparation
  * patients in which cecal intubation was not achieved or scheduled for partial examinations
  * polyps could not be resected due to ongoing anticoagulation or could not be retrieved for pathologic assessment

SUMMARY:
Several reports have suggested that an endoscopic diagnosis of adenoma, by means of narrow band imaging (NBI), might allow the determination of polyp management and surveillance interval, particularly in patients with diminutive polyps (< 5mm), in which the advanced histological features are uncommon and the prevalence of invasive cancer is negligible (1). On this basis, the American Society of Gastrointestinal Endoscopy (ASGE) has set an initiative evaluating the applicability of real-time endoscopic polyp assessment in clinical practice (1), which states that:

1. for diminutive polyps to be resected and discarded without pathologic assessment, endoscopic technology (when used with high confidence) used to determine histology of polyps < 5mm in size, when combined with the histopathologic assessment of polyps >5 mm in size, should provide a > 90% agreement in assignment of post-polypectomy surveillance intervals when compared to decisions based on pathology assessment of all identified polyps.
2. In order for a technology to be used to guide the decision to leave suspected rectosigmoid hyperplastic polyps <5 mm in size in place (without resection), the technology should provide > 90% negative predictive value (when used with high confidence) for adenomatous histology

This strategy could potentially exert a significant impact on colonoscopy practice, by decreasing at some extent pathology-associated costs, although those related to histological analysis of >5mm polyps is maintained.

In a recent study performed in our Centre (2), we restricted the application of the resect and discard strategy to patients with small or diminutive polyps only, achieving an accordance between endoscopy-directed and histology-directed surveillance strategy of about 85% in both populations. This approach, where decisions on patient management are driven only by the "in vivo" endoscopic assessment, provides on one hand a slightly lower accordance than the threshold of 90% set by the PIVI, but on the other one it allows the complete spare of pathology related costs, although for a smaller proportion of patients. Moreover we observed a negative predictive value of 86% for the presence of adenoma within the diminutive polyps cohort, although a separate analysis for left sided ones was not performed.

AIms of this single center, prospective, observational study:

1. To prospectively evaluate the accordance between the endoscopy-directed and histology-directed surveillance strategies by applying the resect and discard strategy for diminutive polyps according to the PIVI statements
2. To assess the economic impact of the resect and discard strategy when applied either according to the PIVI statements or to restrictedly to subjects with diminutive polyps only
3. To provide a temporary validation of diagnostic performances of the resect and discard strategy for our group and the potential presence of a learning effect for the methodology
4. Accordance between endoscopists' and nurses' categorization of adenomas according to standardized criteria (see below)

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy for routine indications (screening, symptoms, surveillance).

Exclusion criteria:

* patients with CRC history or hereditary polyposis syndromes or hereditary non-polyposis colorectal cancer
* patients with inadequate bowel preparation
* patients in which cecal intubation was not achieved or scheduled for partial examinations
* polyps could not be resected due to ongoing anticoagulation or could not be retrieved for pathologic assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult (18-80 yrs) outpatients undergoing colonoscopy for routine indications (screening, symptoms, surveillance).
  Exclusion criteria:
  * patients with CRC history or hereditary polyposis syndromes or hereditary non-polyposis colorectal cancer
  * patients with inadequate bowel preparation
  * patients in which cecal intubation was not achieved or scheduled for partial examinations
  * polyps could not be resected due to ongoing anticoagulation or could not be retrieved for pathologic assessment
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
proportion of cases in which the accordance between the endoscopy-directed and histology-directed surveillance strategies by applying the resect and discard strategy for diminutive polyps according to the PIVI statements was observed | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Valduce, Como, Italy

REFERENCES:
- [Derived] Paggi S, Rondonotti E, Amato A, Fuccio L, Andrealli A, Spinzi G, Radaelli F. Narrow-band imaging in the prediction of surveillance intervals after polypectomy in community practice. Endoscopy. 2015 Sep;47(9):808-14. doi: 10.1055/s-0034-1392042. Epub 2015 Jun 12. PMID 26070008